CLINICAL TRIAL: NCT01535534
Title: Evaluation of Mediators of Inflammation, Prognostic Markers and Genetic Polymorphisms in Patients With Sepsis
Brief Title: Mediators of Inflammation, Prognostic Markers and Genetic Polymorphisms in Patients With Sepsis
Acronym: MaSep
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Universitätsmedizin Mannheim (Other)
Responsible Party: Principal Investigator, Dr. med. Ursula Hoffmann, Principal Investigator, Universitätsmedizin Mannheim
Other Study IDs: 2011-384N-MA
Record Dates: First submitted 2012-02-14; First posted 2012-02-17 (Estimated); Last update posted 2020-08-27 (Actual); Status verified 2020-08

CONDITIONS: Sepsis
Keywords: sepsis; inflammation; diagnosis; prognosis; survival; mortality
MeSH Terms: conditions — Sepsis; Inflammation; Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Peripheral blood samples
Oversight: Data Monitoring Committee: No

SUMMARY:
During the past years many investigators have focused on the immunological changes in sepsis disease, and great attention has been paid to the development of practicable means of immunomonitoring. Little is known about diagnostic and prognostic vascular biomarkers during the time course of patients with sepsis.

DETAILED DESCRIPTION:
Primary Outcome Measures:

New diagnostic and prognostic markers for septic patients

Estimated Enrollment: 300 patients Study Start Date: January 2012 Estimated Study Completion Date: open Estimated Primary Completion Date: open

Intervention Details:

Procedure: vein puncture comparison of different inflammatory markers in the blood of septic patients

ELIGIBILITY:
Inclusion Criteria:

* SIRS-Criteria
* Proven Infection
* One sepsis-induced organ-failure
* Adults < 18 years old

Exclusion Criteria:

* Anemia
* Pregnancy
* Blood donor in the last 3 month

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients suffering from sepsis
Sampling Method: Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2012-01 (Actual); Primary Completion 2018-12 (Actual); Study Completion 2021-12 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Ursula Hoffmann, MD, Principal Investigator — Universitätsmedizin Mannheim; Michael Behnes, MD, Study Director — Universitätsmedizin Mannheim
Locations (1):
- University Medical Centre Mannheim, Mannheim, Baden-Wurttemberg, Germany

REFERENCES:
- [Derived] Hamed S, Behnes M, Pauly D, Lepiorz D, Barre M, Becher T, Lang S, Akin I, Borggrefe M, Bertsch T, Hoffmann U. Diagnostic value of Pentraxin-3 in patients with sepsis and septic shock in accordance with latest sepsis-3 definitions. BMC Infect Dis. 2017 Aug 9;17(1):554. doi: 10.1186/s12879-017-2606-3. PMID 28793880
- [Derived] Behnes M, Bertsch T, Lepiorz D, Lang S, Trinkmann F, Brueckmann M, Borggrefe M, Hoffmann U. Diagnostic and prognostic utility of soluble CD 14 subtype (presepsin) for severe sepsis and septic shock during the first week of intensive care treatment. Crit Care. 2014 Sep 5;18(5):507. doi: 10.1186/s13054-014-0507-z. PMID 25190134